CLINICAL TRIAL: NCT01876160
Title: Analysis of Sensory and Motor Thresholds During Transcutaneous Electrical Stimulation in Different Sexes and Ages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: U1111-1143-6220
Record Dates: First submitted 2013-05-27; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Individuals
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- threshold of sensory perception (Experimental): Eighty healthy volunteers were evaluated; 40 women and 40 men divided into two equal groups of young and elderly subjects. Half of the individuals in each group were stimulated with 5 and 50Hz frequency, with pulse duration of 20, 100, 400, 1000 and 3000µs applied on the flexor muscle bellies of the wrist and fingers. The threshold of sensory perception was identified as the first sensation of increased current intensity and the threshold of motor response as the minimum muscle contraction detected.
  Interventions: Other: Transcutaneous electrical nerve stimulation
- threshold of motor response (Experimental): Eighty healthy volunteers were evaluated; 40 women and 40 men divided into two equal groups of young and elderly subjects. Half of the individuals in each group were stimulated with 5 and 50Hz frequency, with pulse duration of 20, 100, 400, 1000 and 3000µs applied on the flexor muscle bellies of the wrist and fingers. The threshold of motor response as the minimum muscle contraction detected.
  Interventions: Other: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: Transcutaneous electrical nerve stimulation

SUMMARY:
The sensory and motor perception thresholds can influence the therapeutic effects of Transcutaneous Electrical Nerve Stimulation. This study aimed to determine the threshold of sensory perception and the threshold of motor response in young and elderly subjects of both sexes. Eighty healthy volunteers were evaluated; 40 women and 40 men divided into two equal groups of young and elderly subjects. Half of the individuals in each group were stimulated with 5 and 50Hz frequency, with pulse duration of 20, 100, 400, 1000 and 3000µs applied on the flexor muscle bellies of the wrist and fingers. The threshold of sensory perception was identified as the first sensation of increased current intensity and the threshold of motor response as the minimum muscle contraction detected. The results were submitted to ANOVA test, followed by the Tukey test, with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals

Exclusion Criteria:

* not present: previous circulatory, nervous or metabolic diseases, metal implants in areas to be studied; fracture on upper limb studied; history of pain or injury in areas to be studied.
* are not in menstrual period or a week before it
* not be making use of drugs that affect the nervous system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Analysis of sensory thresholds | 1 years
  A pulse generator was used for data collection, with constant current intensity, and the following parameters were used for current stimulation: square biphasic wave, and pulse-width varying in 20, 50, 100, 200,300, 500, 1000 and 3000µs, at a frequency of 5 or 50Hz. During the procedure, the volunteers remained seated, with the forearm in supination, resting on a table. The tests always initiated with 20µs pulse-width, with high intensity until the threshold of sensory perception were reached. At this point, the intensity was reset and the procedure began again, followed by the next pulse duration, progressively evolving up to 3000µs and repeated three times with a 10-minute interval between the tests. The procedures were carried out with a 72 hour minimum interval for different frequencies.
Analysis of Motor thresholds | 1 years
  A pulse generator was used for data collection, with constant current intensity, and the following parameters were used for current stimulation: square biphasic wave, and pulse-width varying in 20, 50, 100, 200,300, 500, 1000 and 3000µs, at a frequency of 5 or 50Hz. During the procedure, the volunteers remained seated, with the forearm in supination, resting on a table. The tests always initiated with 20µs pulse-width, with high intensity until the threshold of motor response were reached. At this point, the intensity was reset and the procedure began again, followed by the next pulse duration, progressively evolving up to 3000µs and repeated three times with a 10-minute interval between the tests. The procedures were carried out with a 72 hour minimum interval for different frequencies.